CLINICAL TRIAL: NCT01166633
Title: A Randomized , Open Label, Dose Titration Study to Evaluate the Effect of Pitavastatin Versus Atorvastatin in Patients With Hypercholesterolemia and Mild to Moderate Hepatic Damage
Brief Title: Efficacy and Safety Study of Pitavastatin Versus Atorvastatin to Treat Hypercholesterolemia
Acronym: PITCH
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: JW Pharmaceutical (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CWP-PTV-707
Record Dates: First submitted 2010-07-19; First posted 2010-07-21 (Estimated); Last update posted 2022-04-11 (Actual); Status verified 2022-04

CONDITIONS: Hypercholesterolemia
Keywords: Hydroxymethylglutaryl-CoA Reductase Inhibitors; hyperlipidemia
MeSH Terms: conditions — Hypercholesterolemia; Hyperlipidemias | interventions — pitavastatin; Atorvastatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Pitavastatin 2 mg (Experimental)
  Interventions: Drug: pitavastatin
- Atorvastatin 10mg (Active Comparator)
  Interventions: Drug: atorvastatin

INTERVENTIONS:
Drug: pitavastatin — pitavastatin 2mg per daily
  Other Names: LIVALO
  Arms: Pitavastatin 2 mg
Drug: atorvastatin — atorvastatin 10mg per daily
  Other Names: LIPITOR
  Arms: Atorvastatin 10mg

SUMMARY:
Statin is an effective drug to treat hyperlipidemia (hypercholesterolemia), and it rarely leads to hepatic damage to the patients with hepatic disorder. For these patients, intensive monitoring is required.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged between 25 and 75
* Patients who signed informed consent forms of their own volition;
* Patients who had taken statins for 2 months and longer or whose fasting LDL-C levels, were 130mg/dL and over (Friedewald's formula);
* Patients whose ALT levels were 1.25 to 2.5 times higher than the upper limit of normal

Exclusion Criteria:

* Patients with uncompensated liver cirrhosis.
* Patients whose total bilirubin levels were over 2 times higher than the upper limit of normal.
* Patients who had taken antiviral drugs for viral hepatitis.
* Patients who experienced cerebrovascular diseases or myocardial infarction within 3 months before screening visit or patients with heart failure (NYHA class IV).
* Patients whose triglyceride(TG) levels were 400mg/dL or higher.
* Patients with uncontrolled hypertension (DBP≧100mmHg)
* Patients under suspicion of renal dysfunction (serum creatinine≧2.0mg/dL)
* Patients whose CK levels were over 2.5 times higher than the upper limit of normal.
* Patients with uncontrolled hypothyroidism although drug treatment (TSH≧ULN×1.5)
* Female patients who were nursing or being pregnant or were planning on becoming pregnant.
* Patients judged to be unsuitable by investigators.

Ages: 25 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2009-06; Primary Completion 2010-11 (Actual); Study Completion 2011-02 (Actual)

PRIMARY OUTCOMES:
Proportion of the subjects whose ALT levels were over CTCAE grade II after treatment | 12 weeks

SECONDARY OUTCOMES:
1.Changes in ALT after treatment | 12 weeks
2.Changes in AST after treatment | 12 weeks
3.Changes in LDL-C, TC, TG and HDL-C after treatment | 12 weeks
4.Changes in fat in liver after treatment | 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Kyoo-Rok Han, Principal Investigator — Kangdong Sacred Heart Hospital